CLINICAL TRIAL: NCT06228560
Title: Multi-center,Randomized,Double-blind Phase II Study to Evaluate the Efficacy and Safety of LP-003 in Patients With Chronic Spontaneous Urticaria (CSU) Who Remain Symptomatic Despite Antihistamine (H1) Treatment
Brief Title: Efficacy and Safety of LP-003 in Patients With CSU Who Remain Symptomatic Despite Antihistamine (H1) Treatment
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Longbio Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: P10-LP003-03
Record Dates: First submitted 2024-01-18; First posted 2024-01-29 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-12

CONDITIONS: Chronic Spontaneous Urticaria
MeSH Terms: conditions — Chronic Urticaria | interventions — Omalizumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- LP-003 group 1 (Experimental): Participants received LP-003 subcutaneously during the 24-week treatment period
  Interventions: Biological: LP-003
- LP-003 group 2 (Experimental): Participants received LP-003 subcutaneously during the 24-week treatment period
  Interventions: Biological: LP-003
- LP-003 group 3 (Experimental): Participants received LP-003 subcutaneously during the 24-week treatment period
  Interventions: Biological: LP-003
- Omalizumab (Active Comparator): Participants received omalizumab 300 mg subcutaneously every 4 weeks during the 24-week treatment period
  Interventions: Biological: Omalizumab
- Placebo (Placebo Comparator): Participants received placebo subcutaneously every 4 weeks during the 24-week treatment period
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: LP-003 — Liquid in vial
  Arms: LP-003 group 1; LP-003 group 2; LP-003 group 3
Biological: Placebo — Liquid in vial
  Arms: Placebo
Biological: Omalizumab — Liquid in vial
  Arms: Omalizumab

SUMMARY:
The study is a Phase II, multicenter, randomized, double-blind study to evaluatethe efficacy and safety of LP-003 administered subcutaneously as an add-on therapy for the treatment of adult patients aged 18-75 who have been diagnosed with refractory CSU and who remain symptomatic despitestandard-dose H1 antihistamine treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18 to 75 years at the screening period.
2. Presence of wheals with itching for ≥ 6 weeks prior to randomization. At the screening visit, subjects had taken double or more than the approved dose, or a combination of two or more H1 antihistamines for the treatment of chronic spontaneous urticaria for at least 2 weeks. Within the 7 days preceding randomization, the Urticaria Activity Score 7 (UAS7) was ≥16 (range 0-42), Itch Severity Score 7 (ISS7) was ≥8 (range 0-21), at least one UAS (range 0-6) was ≥4 on any screening visit day, and there must be a current record of medication use.
3. Subjects must not miss more than one diary record (morning or night) within 7 days prior to randomization (day 1), and are willing and able to complete daily symptom electronic diary records during the study period;
4. Male participants and their partners or female participants must agree to take one or more non pharmacological contraceptive measures (such as complete abstinence, contraceptive ring, partner ligation, etc.) during the trial period and within 6 months after the end of the trial and have no plans for sperm or egg donation.
5. Agree to participate in this clinical trial and voluntarily sign an informed consent form.

Exclusion Criteria:

1. The subject has a primary or sole trigger for chronic urticaria (chronic Induced urticaria), including artificial urticaria (symptomatic skin scratch disease), cold, heat, sun, pressure, delayed pressure, water, cholinergic, or contact urticaria;
2. Other medical conditions accompanied by symptoms of urticaria or angioedema including, but not limited to, urticarial vasculitis, pigmented urticaria, erythema multiforme, mastocytosis, hereditary urticaria, or drug-induced urticaria;
3. Any other dermatologic condition with chronic itching, such as atopic dermatitis, herpetic pemphigoid, herpetic dermatitis, senile itching, or psoriasis, which in the judgment of the Investigator may affect the evaluation of the study and the results of the study;
4. Subjects with clinically significant conditions such as (but not limited to) unstable ischemic heart disease, NYHA Class III/IV left ventricular failure, cardiac arrhythmias, uncontrolled hypertension, cerebrovascular disease, neurodegenerative, or other neurological disorders, uncontrolled hypothyroidism and hyperthyroidism and other autoimmune disorders, hypokalemia, hyper adrenergic state; past diagnosis of malignancy (other than basal cell carcinoma or squamous cell skin cancer); history of myocardial infarction within 12 months prior to screening;
5. Acute active infections requiring treatment at screening, including but not limited to, pulmonary infections, tuberculosis;
6. Positive hepatitis B surface antigen or hepatitis B core antibody (except for HBV-DNA testing below the lower limit of the research center's test) at screening; positive hepatitis C virus antibody, human immunodeficiency virus (HIV) antibody, and anti-syphilis helical antibody (TP-Ab) (except for those who are negative for RPR or TRUST);
7. Clinically significant cardiovascular, neurological, psychiatric, metabolic, hepatic, or other abnormalities identified during the Screening Period that may affect the interpretation of the study results and/or the safety of the subject;
8. Comorbid neurological or psychiatric disorders that prevent or prevent cooperation; patients with disabilities as defined by law (blindness, deafness, mute, mental retardation, psychiatric disorders, etc.);
9. Major surgery within 8 weeks prior to screening or surgery planned during the study period;
10. Evidence of historical or ongoing alcohol or substance abuse in the 6 months prior to screening;
11. Poor compliance, such as low medication adherence, inability to accurately complete a diary card, or use of prohibited medications;
12. Pregnant women, nursing mothers, or those with recent birth plans;
13. Patients who have participated in clinical trials of other drugs within the last 3 months;
14. Those who are considered by the investigator to be unfit to participate in the clinical trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 202 (Actual)
Dates: Start 2024-01-26 (Actual); Primary Completion 2025-04-17 (Actual); Study Completion 2025-11-14 (Actual)

PRIMARY OUTCOMES:
The proportion of participants achieving complete absence of wheals and itching (UAS7 = 0) at week 12 | Week 12

SECONDARY OUTCOMES:
The incidence of adverse events during the study | 40 weeks
The proportion of participants with no hives (HSS7 = 0) at week 4, 8, 12, 16, 20, 24, 32, and 40 | Week 4, 8, 12, 16, 20, 24, 32, and 40
The proportion of participants achieving complete absence of wheals and itching (UAS7 = 0) at week 4, 8, 16, 20, 24, 32, and 40 | Week 4, 8, 16, 20, 24, 32, and 40
The proportion of participants achieving complete absence of angioedema (AAS7 = 0) at week 4, 8, 12, 16, 20, 24, 32, and 40 | Week 4, 8, 12, 16, 20, 24, 32, and 40
The proportion of participants with controlled disease activity (UAS7 ≤ 6) at week 4, 8, 12, 16, 20, 24, 32, and 40 | Week 4, 8, 12, 16, 20, 24, 32, and 40
Change From Baseline in UAS7, HSS7, ISS7, AAS7 at week 4, 8, 12, 16, 20, 24, 32, and 40 | Baseline and week 4, 8, 12, 16, 20, 24, 32, and 40
Change From Baseline in Chronic Urticaria Quality of Life Questionnaire (CU-Q2oL) at week 4, 8, 12, 16, 20, 24, 32, and 40 | Baseline and week 4, 8, 12, 16, 20, 24, 32, and 40
Blood concentrations of LP-003, free IgE, total IgE, anti-drug antibodies (ADA), and neutralizing antibodies (Nab) during the study | 40 weeks

CONTACTS AND LOCATIONS:
Locations (20):
- China (20):
  - Beijing Friendship Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Peking Union Medical College Hospital, Chinese Academy of Medical Sciences, Beijing, Beijing Municipality
  - Peking University Third Hospital, Beijing, Beijing Municipality
  - The First Affiliated Hospital of China Medical University, Beijing, Beijing Municipality
  - The First Hospital of Peking University, Beijing, Beijing Municipality
  - The First Affiliated Hospital of PLA Army Medical University, Chongqing, Chongqing Municipality
  - Fujian Medical University Union Hospital, Fuzhou, Fujian
  - Dermatology Hospital of Southern Medical University, Guangzhou, Guangdong
  - The Second Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong
  - Tongji Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei
  - The Second XiangYa Hospital of Central South University, Changsha, Hunan
  - Hospital of Dermatology, Chinese Academy of Medical Sciences and Peking Union Medical College, Nanjing, Jiangsu
  - Shengjing Hospital of China Medical University, Shenyang, Liaoning
  - Ruijin Hospital Affiliated to Shanghai Jiaotong University School of Medicine, Shanghai, Shanghai Municipality
  - Shanghai Skin Disease Hospital, Shanghai, Shanghai Municipality
  - the Second Affiliated Hospital of Xi'an Jiaotong University, Xi’an, Shanxi
  - Hangzhou First People's Hospital, Hangzhou
  - The Second Affiliated Hospital Zhejiang University School of Medicine, Hangzhou
  - Wuhan NO.1 Hospital, Wuhan
  - Affiliated Hospital of Jiangsu University, Zhenjiang